CLINICAL TRIAL: NCT04062864
Title: Validity of Pupil Diameter for Pain Monitoring During General Anesthesia in Children : a Prospective Observational Study
Brief Title: Pupillometer as a Pain Index During General Anesthesia
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Other Study IDs: 1906-121-1043
Record Dates: First submitted 2019-08-18; First posted 2019-08-20 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Anesthesia, General; Pupil; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pupil size — Measures the diameter of pupil before and after painful stimuli
  Other Names: Pupillometer

SUMMARY:
This study evaluates the validity of pupil diameter as an indicator of pain during surgery under general anesthesia.

DETAILED DESCRIPTION:
Pupil diameter is known to be strongly correlated with sympathetic tone. During surgery under general anesthesia, there is no standardized means of pain assessment. As pain activates sympathetic nervous system, we hypothesized that pupil diameter can be a marker for pain during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing surgery under general anesthesia with total time of less than two hours

Exclusion Criteria:

* Children whose parent or legal guardian declined to enroll
* Any use of opioids during surgery
* History of hypersensitivity to any anesthetic agents
* Any medication that can affect sympathetic nervous activity
* Presence of underlying ophthalmologic disease

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing surgery under general anesthesia at Seoul National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Pupil diameter | From start of anesthesia to end of anesthesia
  Pupil diameter before and after painful stimuli (skin incision, train-of-four stimulation)

SECONDARY OUTCOMES:
Bispectral index | From start of anesthesia to end of anesthesia
  Bispectral index before and after painful stimuli (skin incision, train-of-four stimulation)
Pleth variability index | From start of anesthesia to end of anesthesia
  Pleth variability index before and after painful stimuli (skin incision, train-of-four stimulation)

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- SNUH, Seoul, Jongno Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aissou M, Snauwaert A, Dupuis C, Atchabahian A, Aubrun F, Beaussier M. Objective assessment of the immediate postoperative analgesia using pupillary reflex measurement: a prospective and observational study. Anesthesiology. 2012 May;116(5):1006-12. doi: 10.1097/ALN.0b013e318251d1fb. PMID 22446982
- [Background] Barvais L, Engelman E, Eba JM, Coussaert E, Cantraine F, Kenny GN. Effect site concentrations of remifentanil and pupil response to noxious stimulation. Br J Anaesth. 2003 Sep;91(3):347-52. doi: 10.1093/bja/aeg178. PMID 12925472
- [Background] Hofle M, Kenntner-Mabiala R, Pauli P, Alpers GW. You can see pain in the eye: pupillometry as an index of pain intensity under different luminance conditions. Int J Psychophysiol. 2008 Dec;70(3):171-5. doi: 10.1016/j.ijpsycho.2008.06.008. Epub 2008 Jun 28. PMID 18644409
- [Background] Julien-Marsollier F, Rachdi K, Caballero MJ, Ayanmanesh F, Vacher T, Horlin AL, Skhiri A, Brasher C, Michelet D, Dahmani S. Evaluation of the analgesia nociception index for monitoring intraoperative analgesia in children. Br J Anaesth. 2018 Aug;121(2):462-468. doi: 10.1016/j.bja.2018.03.034. Epub 2018 Jun 5. PMID 30032886
- [Background] Kaye AD, Fox CJ, Padnos IW, Ehrhardt KP Jr, Diaz JH, Cornett EM, Chandler D, Sen S, Patil S. Pharmacologic Considerations of Anesthetic Agents in Pediatric Patients: A Comprehensive Review. Anesthesiol Clin. 2017 Jun;35(2):e73-e94. doi: 10.1016/j.anclin.2017.01.012. Epub 2017 Apr 14. PMID 28526162
- [Background] Mulier J, Dekock M. Opioid free general anesthesia, a new paradigm? Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):441-443. doi: 10.1016/j.bpa.2017.11.005. Epub 2017 Dec 6. No abstract available. PMID 29739534
- [Background] Muller MP, Tomlinson G, Marrie TJ, Tang P, McGeer A, Low DE, Detsky AS, Gold WL. Can routine laboratory tests discriminate between severe acute respiratory syndrome and other causes of community-acquired pneumonia? Clin Infect Dis. 2005 Apr 15;40(8):1079-86. doi: 10.1086/428577. Epub 2005 Mar 16. PMID 15791504
- [Background] Paulus J, Roquilly A, Beloeil H, Theraud J, Asehnoune K, Lejus C. Pupillary reflex measurement predicts insufficient analgesia before endotracheal suctioning in critically ill patients. Crit Care. 2013 Jul 24;17(4):R161. doi: 10.1186/cc12840. PMID 23883683
- [Background] Sabourdin N, Barrois J, Louvet N, Rigouzzo A, Guye ML, Dadure C, Constant I. Pupillometry-guided Intraoperative Remifentanil Administration versus Standard Practice Influences Opioid Use: A Randomized Study. Anesthesiology. 2017 Aug;127(2):284-292. doi: 10.1097/ALN.0000000000001705. PMID 28719527
- [Background] Silins V, Brasher C, Antus F, Michelet D, Hilly J, Grace R, Dahmani S. Predicting postoperative morphine consumption in children. Anaesth Crit Care Pain Med. 2017 Jun;36(3):179-184. doi: 10.1016/j.accpm.2016.08.005. Epub 2016 Oct 4. PMID 27717898
- [Background] Sultana A, Torres D, Schumann R. Special indications for Opioid Free Anaesthesia and Analgesia, patient and procedure related: Including obesity, sleep apnoea, chronic obstructive pulmonary disease, complex regional pain syndromes, opioid addiction and cancer surgery. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):547-560. doi: 10.1016/j.bpa.2017.11.002. Epub 2017 Nov 16. PMID 29739543
- [Background] Urban BW, Bleckwenn M. Concepts and correlations relevant to general anaesthesia. Br J Anaesth. 2002 Jul;89(1):3-16. doi: 10.1093/bja/aef164. No abstract available. PMID 12173238
- [Background] Wessel DL. Hemodynamic responses to perioperative pain and stress in infants. Crit Care Med. 1993 Sep;21(9 Suppl):S361-2. doi: 10.1097/00003246-199309001-00037. No abstract available. PMID 8365227
- [Background] Wildemeersch D, Peeters N, Saldien V, Vercauteren M, Hans G. Pain assessment by pupil dilation reflex in response to noxious stimulation in anaesthetized adults. Acta Anaesthesiol Scand. 2018 Sep;62(8):1050-1056. doi: 10.1111/aas.13129. Epub 2018 Apr 19. PMID 29671874
- [Background] Won YJ, Lim BG, Kim YS, Lee M, Kim H. Usefulness of surgical pleth index-guided analgesia during general anesthesia: a systematic review and meta-analysis of randomized controlled trials. J Int Med Res. 2018 Nov;46(11):4386-4398. doi: 10.1177/0300060518796749. Epub 2018 Sep 9. PMID 30198405